CLINICAL TRIAL: NCT06693167
Title: Adjuvant Treatment of Postoperative Pain Following Endoscopic Carpal Tunnel Surgery by Auriculotherapy
Acronym: AURDO1
Status: Completed | Type: Observational
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Other Study IDs: 0990-0279
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Chirurgical Intervention; Auriculotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: chirurgie canal carpien — study compares a group of patients who received a preoperative auriculotherapy session followed by standard analgesic treatment to a group who received only standard analgesic treatment, and this, during the three days following surgery (D1, D2, and D3).

SUMMARY:
Retrospective study on the effect of auriculotherapy on postoperative pain after carpal tunnel surgery

DETAILED DESCRIPTION:
the project consists of a retrospective analysis of data from the medical records of patients followed by Doctor, between 2016 and 2017, at the Bizet Clinic. This study includes measurements of pain levels and analgesic consumption in patients who received during their care in the clinic a preoperative auriculotherapy session offered by the clinic, during the three days following carpal tunnel surgery. For comparison, this studie also includes a group who underwent the same surgery treated only with analgesics. The objective of study is to analyze the results obtained in the two groups in order to evaluate the effectiveness of auriculotherapy for the management of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 84 years.
* Patients suffering from carpal tunnel syndrome for whom elective endoscopic surgery is indicated

Exclusion Criteria:

* Have already benefited from an auriculotherapy session.
* Presence of cryoglobulinemia.
* Presence of Raynaud's syndrome.
* Presence of hemoglobinopathy (hemoglobin and capillary abnormalities).
* Allergy to cold.
* Presence of dermatological lesions on the auricle of one of the two ears

Ages: 18 Years to 84 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from carpal tunnel syndrome for whom elective endoscopic surgery is indicated
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
demonstrate the effectiveness of auriculotherapy in the management of postoperative pain | Day1, Day2 and Day 3
  pain assessment scale

SECONDARY OUTCOMES:
reducing the consumption of painkillers | Day1, Day2 and Day 3
  number of tablets in grams

REFERENCES:
- See also: 6- Sator-Katzenschlager, S. M., Scharbert, G., Kozek-Langenecker, S. A., Dolezal, S., Michalek-Sauberer, A., Kress, H. G., & Heinze, G. (2003). The short- and long-term benefit in chronic low back pain through adjuvant electrical versus manual auricular — https://pubmed.ncbi.nlm.nih.gov/15105215/